CLINICAL TRIAL: NCT06151665
Title: A Comparative Study Between Single Rotary File System and Conventional Manual K-File in Pulpectomy of Primary Molars.
Brief Title: Single Rotary File System Versus Conventional Manual K-file in Pulpectomy of Primary Molars.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah magdy, assistant lecturer of pediatric dentistry, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PED23-3D
Record Dates: First submitted 2023-11-16; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Endodontically Treated Teeth
Keywords: primary-molars; pulpectomy; Rotary
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Intervention Model Description: Primary molars with irreversible pulpitis
Who Masked: Outcomes Assessor
Masking Description: an external pediatric Dentist will assess the radiographic and clinical follow-up of the enrolled patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Rotary file (Experimental): single rotary file will be used in primary molars to preform pulpectomy then restored with zinc oxide eugenol and stainless steel crown.
  Interventions: Procedure: single file rotary
- Conventional Manual Files (Active Comparator): Conventional Manual Stainless steel K files will be used in primary molars to preform pulpectomy then restored with zinc oxide eugenol and stainless steel crown.
  Interventions: Procedure: Conventional Manual K files

INTERVENTIONS:
Procedure: single file rotary — Kedo-S plus file is the fifth generation of pediatric files will be used in pulpectomy of primary molars
  Arms: Single Rotary file
Procedure: Conventional Manual K files — Stainless-steel K files is the golden standard files used in pulpectomy of primary molars
  Arms: Conventional Manual Files

SUMMARY:
The sample size will be divided between two groups, Group A pulpectomy will be done using single rotary file in primary molars and group B pulpectomy will be done using manual K file system. follow up of the patients and clinical and radiographical success rates of cases will be seen.

DETAILED DESCRIPTION:
Each patient will have access in the primary molar and pulpectomy procedure will be done according to inclusion and exclusion criteria , the patients will be divided according to two groups Group A using single File rotary and group B manual K file system. Time will be recorded in each procedure and each patient will receive stainless steel crown. Follow up for the patients will be done clinical and radiographical success will be seen, postoperative pain will be measured and all data will be collected and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Absence of external or internal root resorption
2. presence of two thirds of the root
3. Primary molars with deep caries and irreversible pulpitis that require pulpectomy in a single visit. Molars can be vital with a history of spontaneous pain or non-vital as indicated by absence of bleeding from the pulp.

Exclusion Criteria:

* Children with physical, intellectual disability or medical conditions that may complicate treatment.
* Teeth with poor prognosis due to the presence of a sinus, excessive mobility or advanced bone resorption.
* Teeth with radiolucent areas in furcation regions.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and Radiographical Success | 1 year
  Clinical evaluation to swelling, fistula and pain on percussion by clinical examination followed by a radiographic evaluation to absence of periapical and inter-radicular radiolucency, external or internal root resorption according to radiographic images

SECONDARY OUTCOMES:
postoperative pain | 3 days
  Postoperative pain will be recorded at six, 12, 24, 48, and72 hours following the pulpectomy. To ensure standardization, the same parent will be asked to record the pain intensity at all intervals as told by the child. Wong Bakers FACES Pain Rating Scale (WB-FPRS) will be employed to assess post-operative pain. The scale is a pictorial representation of the discomfort level experienced by children which comprise six faces, each depicting an expression of pain. Also visual Analogue Scale (VAS) for pain assessment will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jeevanandan G, Govindaraju L. Clinical comparison of Kedo-S paediatric rotary files vs manual instrumentation for root canal preparation in primary molars: a double blinded randomised clinical trial. Eur Arch Paediatr Dent. 2018 Aug;19(4):273-278. doi: 10.1007/s40368-018-0356-6. Epub 2018 Jul 12. PMID 30003514
- [Background] Panchal V, Jeevanandan G, Subramanian E. Comparison of instrumentation time and obturation quality between hand K-file, H-files, and rotary Kedo-S in root canal treatment of primary teeth: A randomized controlled trial. J Indian Soc Pedod Prev Dent. 2019 Jan-Mar;37(1):75-79. doi: 10.4103/JISPPD.JISPPD_72_18. PMID 30804311
- [Background] Priyadarshini P, Jeevanandan G, Govindaraju L, Subramanian EMG. Clinical evaluation of instrumentation time and quality of obturation using paediatric hand and rotary file systems with conventional hand K-files for pulpectomy in primary mandibular molars: a double-blinded randomized controlled trial. Eur Arch Paediatr Dent. 2020 Dec;21(6):693-701. doi: 10.1007/s40368-020-00518-w. Epub 2020 Mar 17. PMID 32185634
- [Background] Coll JA, Sadrian R. Predicting pulpectomy success and its relationship to exfoliation and succedaneous dentition. Pediatr Dent. 1996 Jan-Feb;18(1):57-63. PMID 8668572